CLINICAL TRIAL: NCT03846570
Title: Formoterol-beclomethasone in Patients With Bronchiectasis: a Randomized Controlled Trial
Acronym: FORZA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient inclusion rate (due to COVID-19 pandemic)
Sponsor: Erasmus Medical Center (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, Menno M. van der Eerden, Pulmonary physician, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL61630.078.18
Record Dates: First submitted 2019-02-14; First posted 2019-02-19 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Bronchiectasis
Keywords: Randomized Controlled Trial; Inhaled corticosteroids; Placebo; Cough
MeSH Terms: conditions — Bronchiectasis; Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Formoterol-beclomethasone (Active Comparator): Formoterol (fumarate dehydrate) 12 microg - beclomethasone (dipropionate) 200 microg administered BID, per inhalation using '100/6' Metered Dose Inhaler.
  Interventions: Drug: Formoterol-beclomethasone
- Placebo (Placebo Comparator): Matching placebo (identically package) administered BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Formoterol-beclomethasone — formoterol (fumarate dihydrate) 12 microg - beclomethasone (dipropionate) 200 microg administered BID, per inhalation using '100/6' Metered Dose Inhaler
  Arms: Formoterol-beclomethasone
Drug: Placebo — Matching placebo (identically package) administered BID
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled study comparing formoterol-beclometason 12/200 mcg BID versus placebo to evaluate the clinical effect on coughing in patients with non-cystic fibrosis (non-CF) bronchiectasis, native to inhaled corticosteroid (ICS) therapy and no history of asthma or chronic obstructive pulmonary disease (COPD)

DETAILED DESCRIPTION:
In the management of non-CF bronchiectasis, bronchodilator treatment (LABA)and use of inhaled corticosteroids (ICS) is still a matter of debate. Previous studies have claimed beneficial effects of ICS (with or without bronchodilator), such as improvement of the HRQL, a reduction in daily sputum volume and/or exacerbation frequency. However, in all previous studies there was no clear exclusion of patients with asthma or COPD, or no use of placebo. The current study will be the first study evaluating the effect of ICS/LABA treatment in non-CF bronchiectasis excluding patients with asthma and COPD.

This is a prospective double-blind randomized controlled trial comparing Formoterol-beclomethasone 12/200 mcg BID versus placebo to evaluate the reduction in cough measured by the Leicester cough questionnaire. Secondary objectives are the improvement of health-related quality of life and symptoms, reduction in sputum production, pulmonary function (FEV1) and the frequency of exacerbation. Furthemore, we will assess the inflammatory response in serum and sputum.

After a wash-out period of 1 month, eligible subjects will be randomized to treatment with formoterol-beclomethasone or matching placebo. All subjects will be treated with the regimen of medication for 3 months. An end-of-study (EOS) visit will be performed after completion of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patient (wheezing, cough and dyspnoea);
* Proven and documented diagnosis of BE by high resolution computed tomography ;
* Stable pulmonary status as indicated by FEV1 (percent of predicted) ≥30%
* Stable clinically phase (ie, subjects free from acute exacerbation for at least 6 weeks prior to the start of the study);
* Stable regimen of standard treatment as chronic treatment for BE, at least for the past 4 weeks prior to screening. And/or macrolides if used as chronic treatment for BE at least for the past 6 months prior to screening;
* Coughing on the majority of days for more than 8 weeks;
* Ability to follow the inhaler device instructions;
* Ability to complete questionnaires;
* Written informed consent.

Exclusion Criteria:

* Possible asthma according to the definition of the Global Initiative for Asthma (GINA);
* Positive histamine provocation test
* Known intolerance for ICS or LABA;
* Women who are pregnant, lactating, or in whom pregnancy cannot be excluded;
* Expected to die within 72 hours after enrolment;
* Cigarette smoking history of > 10 pack-years or current smokers;
* Other cardiopulmonary conditions (other than bronchiectasis) that could modify spirometric values.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Clinical effect on coughing | 3 months
  Using the Leicester Cough Questionnaire (LCQ) at baseline and 3 months. The LCQ is a valid, repeatable 19 item self-completed quality of life measure of chronic cough which is responsive to change. Score range: 19-133 (Higher values represent a better outcome.)

SECONDARY OUTCOMES:
Quality of life in patient with bronchiectasis | 3 months
  Mean Change From Baseline in Patient Reported Outcome Quality of Life Questionnaire for Bronchiectasis (QoL-B) Respiratory Symptoms Domain Score (measured at baseline and 3 months).
  The QoL-B was a disease-specific questionnaire developed for non-Cystic fibrosis Bronchiectasis. It covers 8 dimensions: physical functioning, role functioning, emotional functioning, social functioning, vitality, treatment burden, health perceptions, and respiratory symptoms. Each dimension was scored separately on a scale of 0 to 100, and higher scores represent better outcomes. For this outcome measure, the respiratory symptoms domain score was reported.
Pulmonary function | 3 months
  Spirometry: FEV1
Exacerbation frequency | 3 months
  The frequency of exacerbation requiring an intervention with systemic antibiotics (oral/intravenous [i.v.])
Sputum production | 3 months
  in mL
Dyspnea score | 3 months
  mMRC (Modified Medical Research Council) Dyspnea Scale. This stratifies severity of dyspnea in respiratory diseases.
  Grading from 0 to 4, respectively from 'no dyspnea' to 'very severe dyspnea'.
Incidence of Adverse Events [Safety and Tolerability]). | 3 months
  Incidence of Adverse Events [Safety and Tolerability]).
Sputum culture | 3 months
  Micro organisms isolated during study

OTHER OUTCOMES:
Inflammatory response in serum: C-reactive protein | 3 months
  Measuring high-sensitivity C-reactive protein (mg/L) at baseline and 3 months
Inflammatory response in serum: erythrocyte sedimentation rate | 3 months
  Measuring the erythrocyte sedimentation rate (mm/h) at baseline and 3 months
Inflammatory response in serum: WBC | 3 months
  Measuring the white blood cell (WBC) count including polymorphonuclear leukocytes (10^9/L), neutrophils (10^9/L) and eosinophils (10^9/L) at baseline and 3 months
Inflammatory response in serum: pulmonary type 2 innate lymphoid cells | 3 months
  Measuring pulmonary type 2 innate lymphoid cells including IL-4, IL-5 and IL-13 (all in pg/ml) at baseline and 3 months
Inflammatory response in sputum | 3 months
  Measuring the numbers of pulmonary type 2 innate lymphoid cells (ILC2) per ml sputum, observing any change from baseline to 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Menno M Van der Eerden, Principal Investigator — Erasmus Medical Center; Tjeerd Van der Veer, Principal Investigator — Erasmus Medical Center
Locations (3):
- Netherlands (3):
  - Tjeerd van der Veer, Rotterdam
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - HagaZiekenhuis, The Hague

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 36 months after publication
Access Criteria: Data can be requested immediately following publication up to 36 months, after which the data will be filed in the Erasmus MC respiratory medicine department archives without further research support. Data requests are to be addressed to: research.longziekten@erasmusmc.nl